CLINICAL TRIAL: NCT03200028
Title: CCTAP: Cognitive Control Training for Treatment of AUD-PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Posit Science Corporation (Industry)
Collaborators: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSC-0613-17
Record Dates: First submitted 2017-06-21; First posted 2017-06-27 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Alcohol Use Disorder; Post Traumatic Stress Disorder
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Treatment (Experimental): Computerized plasticity-based adaptive cognitive training requiring a total maximum of 30 treatment sessions, up to 5 sessions per week, 30 minutes per session.
  Interventions: Other: Computerized Plasticity-Based Adaptive Cognitive Training

INTERVENTIONS:
Other: Computerized Plasticity-Based Adaptive Cognitive Training — Thirty minutes of training on computerized exercises that targets executive function, memory and attention.

SUMMARY:
The primary objective of this study is to evaluate the feasibility of the revised brain training program with individuals diagnosed with Alcohol Use Disorder (AUD) and Post-Traumatic Stress Disorder (PTSD).

ELIGIBILITY:
Inclusion Criteria:

* Participant is a Veteran and is enrolled in outpatient Substance Use Disorder treatment within Veteran Affairs Palo Alto Health Care System
* Participant meets Diagnostic and Statistical Manual of Mental Disorders-5 criteria for current Alcohol Use Disorder and seeking treatment for Alcohol Use Disorder
* Participant meets Meet Diagnostic and Statistical Manual of Mental Disorders-5 criteria for current PTSD
* Participant must be willing to perform daily home-based computer exercises for 6 weeks
* Participant must demonstrate mild cognitive deficit on neuropsychological tests at the screening visit
* Participant must be a fluent English speaker from the age of 12
* Participant must have adequate sensorimotor capacity to perform the program, including visual capacity adequate to read from a iPad screen at a normal viewing distance, auditory capacity adequate to understand normal speech, and motor capacity adequate to control a touchpad

Exclusion Criteria:

* Participant with diagnosis of an illness or condition with known cognitive consequences (e.g., schizophrenia, bipolar disorder, cancer, multiple sclerosis, Traumatic Brain Injury, mental retardation or pervasive developmental disorder, epilepsy, Parkinson's Disease, delirium or dementia)
* Participant with active suicidal ideations as measured by the Columbia-Suicide Severity Rating Scale (C-SSRS)
* Participant with problems performing assessments or comprehending or following spoken instructions
* Participant who has been treated within 5 years of the date of consent with a computer-based cognitive training program manufactured by Posit Science
* Participant with current severe traumatic brain injury
* Participant with any type of dementia
* Participant with any type of mental retardation
* Participant with limited ability to speak/read/write/understand English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Acceptability | At 6 weeks
  Acceptability will be evaluated through Cognitive Training Acceptability Measure. This measure is comprised of 17 statements about their training experience and participants will be asked to rate each statement on a 7-point Likert scale from Strongly Disagree to Strongly Agree.
Usability | At 6 weeks
  Usability will be evaluated through the Computer System Usability Questionnaire and System Usability Scale. The Computer System Usability Questionnaire and System Usability Scale is comprised of a total of 29 statements and participants will be asked to rate the usability of the system on a 7-point Likert scale from Strongly Disagree to Strongly Agree.

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Kyu Lee, PhD, Principal Investigator — Posit Science Corporation
Locations (1):
- Veterans Affairs Palo Alto Health Care System, Palo Alto, California, United States